CLINICAL TRIAL: NCT02388282
Title: A New Method for Estimating Dynamic Positive End-expiratory Pressure. Description and Validation With PEEPi Dyn Measured With Transdiaphragmatic Pressure
Brief Title: A New Method for Estimating Dynamic Intrinsic PEEP
Acronym: echoPEEPi
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, dr. Stefano Nava, MD, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Other Study IDs: 7/2015/O/Sper
Record Dates: First submitted 2015-03-09; First posted 2015-03-17 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-08

CONDITIONS: PEEP, Intrinsic; PEEP, Occult; Respiratory Insufficiency
Keywords: dynamic intrinsic PEEP; diaphragm echography; respiratory mechanics
MeSH Terms: conditions — Positive-Pressure Respiration, Intrinsic; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: diaphragm ecography — recording of diaphragm ecography

SUMMARY:
Dinamic intrinsic PEEP is

DETAILED DESCRIPTION:
Dynamic intrinsic positive end-expiratory pressure (PEEPi dyn) play an important pathophysiology role in many acute respiratory pathologies.

The most accurate method to quantify PEEPi dyn is to measure the rise in transdiaphragmatic pressure (Pdi) at end expiration at the point of the contraction of the inspiratory muscles until inspiratory flow starts.

Such method, however, is invasive, poor comfortable and require patient active collaboration.

The purpose of this study is describe a new non-invasive method for estimate PEEPi dyn and validate this method with gold-standard-one.

ELIGIBILITY:
Inclusion Criteria:

* Acute or chronic respiratory failure
* Age >=18 y

Exclusion Criteria:

* Lack of informed consent
* Controindication to the placement of oesophageal and gastric catheter:

esophageal varices, gastric or oesophageal bleeding in the previous 30 days, gastric or oesophageal surgery in the preceding year.

* Cardiac arrest
* Severe emodinamic instability (> 1 vasoacttive drug)
* Acute coronary syndrome (AMI/UA)
* Inability to protect airway
* Respiratory arrest
* Pregnancy suspected or confirmed
* Diaphragm palsy
* Curarization in the preceding five hours
* Mechanical ventilation in controlled mode.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with both acute or chronic respiratory insufficiency, who required respiratory mechanics measurements for clinical purpose.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Correlation and agreement between AutoPEEP recorded with the transdiaphragmatic pressure (Pdi) vs ecography measurements. | 20 minutes

SECONDARY OUTCOMES:
Correlation and agreement between neural inspiratory time and ecographic inspiratory time | 10 minutes
Inter-rater agreement to assest method reliability | 10 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Sant'Orsola Malpighi, Bologna, Italy

REFERENCES:
- [Derived] Bernardi E, Pisani L, Fasano L, Lauria G, Comellini V, Appendini L, Conti G, Tosello F, Pizzolato E, Nava S. A New Ultrasound Method for Estimating Dynamic Intrinsic Positive Airway Pressure: A Prospective Clinical Trial. Am J Respir Crit Care Med. 2018 Aug 1;198(3):392-396. doi: 10.1164/rccm.201706-1292LE. No abstract available. PMID 29558160